CLINICAL TRIAL: NCT00125229
Title: Cerebral Hemodynamic Effects of Hypertonic Solutions in Severely Head-Injured Patients
Status: Terminated | Type: Observational
Why Stopped: Dr. Hladky died Sept 2006 prior to study completion
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: 045-1503-266
Record Dates: First submitted 2005-07-27; First posted 2005-07-29 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Traumatic Brain Injury; Intracranial Hypertension
Keywords: Hypertonic Saline; Mannitol; Intracranial hypertension; Cerebral blood flow; Traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hypertension | interventions — Mannitol; Saline Solution, Hypertonic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: Mannitol
Drug: Hypertonic Saline

SUMMARY:
This is a clinical study comparing the physiologic effects of two hypertonic solutions (mannitol, hypertonic saline) with a particular emphasis on changes in cerebral blood flow in patients with intracranial hypertension following serious traumatic brain injury (TBI).

DETAILED DESCRIPTION:
This is a study comparing effects of two hypertonic solutions (mannitol, 6.4% hypertonic saline) on intracranial hypertension, cerebral blood flow, serum/urine osmolarity in patients with increased intracranial pressure caused by traumatic brain injury. The study is conducted during first 72 hours after the injury without any interference with standard medical treatment as performed at the institution. When the hypertonic solution is indicated by caregiver, the study team is informed and performs a set of physiologic bedside measurements including evaluation of cerebral blood flow and changes in plasma and urine osmolarity. The study is noninvasive and the study protocol does not hamper, in any way, standard care of treatment for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe TBI (motor Glasgow Coma Scale [GCS] score < 5)
* Age > 18 years
* Health care provider indicated a treatment of intracranial hypertension using hyperosmotic agent

Exclusion Criteria:

* Brain dead (GCS 3, fixed dilated pupils)
* Life-threatening systemic injuries (AIS > 4 in an organ system other than brain); AIS = Abbreviated Injury Score
* Hypotension not responsive to fluid resuscitation and low doses of dopamine
* Clinical or imaging sign/suspicion for internal carotid artery injury

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe TBI (motor Glasgow Coma Scale [GCS] score < 5)
  * Age > 18 years
  * Health care provider indicated a treatment of intracranial hypertension using hyperosmotic agent
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2005-08; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hlatky, M.D., Principal Investigator — Center for Neurosurgical Sciences - UTHSC San Antonio
Locations (1):
- Center for Neurosurgery Sciences - UTHSCSA - Surgical Intensive Care Unit (SICU), San Antonio, Texas, United States

REFERENCES:
- [Background] Miller JD, Becker DP, Ward JD, Sullivan HG, Adams WE, Rosner MJ. Significance of intracranial hypertension in severe head injury. J Neurosurg. 1977 Oct;47(4):503-16. doi: 10.3171/jns.1977.47.4.0503. PMID 903804
- [Background] Doyle JA, Davis DP, Hoyt DB. The use of hypertonic saline in the treatment of traumatic brain injury. J Trauma. 2001 Feb;50(2):367-83. doi: 10.1097/00005373-200102000-00030. No abstract available. PMID 11242309
- [Background] Wade CE, Kramer GC, Grady JJ, Fabian TC, Younes RN. Efficacy of hypertonic 7.5% saline and 6% dextran-70 in treating trauma: a meta-analysis of controlled clinical studies. Surgery. 1997 Sep;122(3):609-16. doi: 10.1016/s0039-6060(97)90135-5. PMID 9308620
- [Background] Valadka AB, Robertson CS. Should we be using hypertonic saline to treat intracranial hypertension? Crit Care Med. 2000 Apr;28(4):1245-6. doi: 10.1097/00003246-200004000-00069. No abstract available. PMID 10809326
- [Background] Berger S, Schurer L, Hartl R, Deisbock T, Dautermann C, Murr R, Messmer K, Baethmann A. 7.2% NaCl/10% dextran 60 versus 20% mannitol for treatment of intracranial hypertension. Acta Neurochir Suppl (Wien). 1994;60:494-8. doi: 10.1007/978-3-7091-9334-1_135. PMID 7526628
- [Background] Worthley LI, Cooper DJ, Jones N. Treatment of resistant intracranial hypertension with hypertonic saline. Report of two cases. J Neurosurg. 1988 Mar;68(3):478-81. doi: 10.3171/jns.1988.68.3.0478. PMID 3343621
- [Background] Qureshi AI, Suarez JI, Bhardwaj A, Mirski M, Schnitzer MS, Hanley DF, Ulatowski JA. Use of hypertonic (3%) saline/acetate infusion in the treatment of cerebral edema: Effect on intracranial pressure and lateral displacement of the brain. Crit Care Med. 1998 Mar;26(3):440-6. doi: 10.1097/00003246-199803000-00011. PMID 9504569
- [Background] Qureshi AI, Wilson DA, Traystman RJ. Treatment of elevated intracranial pressure in experimental intracerebral hemorrhage: comparison between mannitol and hypertonic saline. Neurosurgery. 1999 May;44(5):1055-63; discussion 1063-4. doi: 10.1097/00006123-199905000-00064. PMID 10232539
- [Background] Vialet R, Albanese J, Thomachot L, Antonini F, Bourgouin A, Alliez B, Martin C. Isovolume hypertonic solutes (sodium chloride or mannitol) in the treatment of refractory posttraumatic intracranial hypertension: 2 mL/kg 7.5% saline is more effective than 2 mL/kg 20% mannitol. Crit Care Med. 2003 Jun;31(6):1683-7. doi: 10.1097/01.CCM.0000063268.91710.DF. PMID 12794404
- [Background] Battison C, Andrews PJ, Graham C, Petty T. Randomized, controlled trial on the effect of a 20% mannitol solution and a 7.5% saline/6% dextran solution on increased intracranial pressure after brain injury. Crit Care Med. 2005 Jan;33(1):196-202; discussion 257-8. doi: 10.1097/01.ccm.0000150269.65485.a6. PMID 15644669
- [Background] Cruz J, Minoja G, Okuchi K, Facco E. Successful use of the new high-dose mannitol treatment in patients with Glasgow Coma Scale scores of 3 and bilateral abnormal pupillary widening: a randomized trial. J Neurosurg. 2004 Mar;100(3):376-83. doi: 10.3171/jns.2004.100.3.0376. PMID 15035271
- [Background] Tseng MY, Al-Rawi PG, Pickard JD, Rasulo FA, Kirkpatrick PJ. Effect of hypertonic saline on cerebral blood flow in poor-grade patients with subarachnoid hemorrhage. Stroke. 2003 Jun;34(6):1389-96. doi: 10.1161/01.STR.0000071526.45277.44. Epub 2003 May 1. PMID 12730557